CLINICAL TRIAL: NCT00436397
Title: Evaluation of the Radionics Body Localizer System and XPLAN/IMRT for Extra-Cranial Sites: A Pilot Study
Brief Title: A New Radiation Therapy Planning System in Patients Undergoing Radiation Therapy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000304713; P30CA006927 (NIH); FCCC-02604
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: A new radiation therapy planning system may help doctors plan better treatment for patients with cancer.

PURPOSE: This clinical trial is studying a new radiation therapy planning system in patients undergoing radiation therapy for extracranial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of the Radionics Body System™ to immobilize and re-localize patients receiving radiotherapy to extra-cranial sites of cancer.
* Determine the accuracy of radiation dose calculations for extra-cranial sites of cancer when using the XPLAN™-intensity modulated radiation therapy (XPLAN™/IMRT) integrated software in this system.

OUTLINE: Patients receiving radiotherapy have a Body Localizer cast constructed and undergo a CT scan while immobilized in the Body Localizer. Patients undergo another CT scan in the treatment position using the standard alpha cradle. The XPLAN™-intensity modulated radiation therapy (XPLAN™/IMRT)-generated treatment plan is compared to the standard treatment plan to verify that the calculated dose is within 2-3 percent of the planned dose using standard technique. Patients undergo sets of CT scans 3 additional times over the next few weeks for a total of 8 CT scans Patients may undergo additional CT scans before and after radiotherapy treatments for a maximum of 5 CT scans per week performed over the course of radiotherapy.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cancer for which a course of radiotherapy to an extra-cranial site is required

  * Head and neck sites excluded
* Initial treatment field (or cone down field) must be no greater than 12 X 10 cm

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No right heart insufficiency

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Weight must not exceed 150 kilograms (330 pounds)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-06; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Seigenberg, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States